CLINICAL TRIAL: NCT02245152
Title: The Effect of Integrated Prevention and Treatment on Child Malnutrition and Health in Burkina Faso: a Cluster Randomized Intervention Study
Acronym: PROMIS-BF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Helen Keller International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IFPRI-2014-001; DFATD (Other Grant/Funding Number: 52308/5252/0200)
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2017-03

CONDITIONS: Child Acute Malnutrition
Keywords: child acute malnutrition; prevention; behavior change communication; lipid-based nutrient supplement; screening coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROMIS intervention (Experimental): * Small group behavior change communication (BCC) on Essential Nutrition Actions (ENA), Infant and Young Child Feeding (IYCF) and Water, sanitation and hygiene (WASH) is provided during monthly well-baby visits for children 0-17 months of age
  * Caregivers with children 0-17 months of age that attend the well-baby visit will be provided with a monthly dose of LNS (20g/day)
  Interventions: Dietary Supplement: LNS; Behavioral: Child's health and nutrition topics; Behavioral: National policy well-baby visits
- control (Active Comparator): Monthly well-baby visits as prescribed by national policy This arm is the basic comparison arm. Caregivers are invited to frequent the health center once a month for well-baby visits. During these visits necessary vaccinations are administered, child growth and nutrition status is evaluated and preventive counseling on child nutrition and health is provided in large groups of caregivers.
  Interventions: Behavioral: National policy well-baby visits

INTERVENTIONS:
Dietary Supplement: LNS — A monthly dose of LNS (31 sachets of 20g) will be distributed to mothers attending well-baby visits and participating in small group counseling
  Other Names: Lipid-based nutrient supplement (LNS)
  Arms: PROMIS intervention
Behavioral: Child's health and nutrition topics — After the well-baby visit. Caregivers will be invited to participate in a small group counseling or BCC (2-3 caregivers at a time).
  Every month a set of topics related to child's health and nutrition will be treated. These BCC sessions will be organized in an interactive way centering around the condition of the participating children.
  Arms: PROMIS intervention
Behavioral: National policy well-baby visits

SUMMARY:
Globally, child undernutrition is the underlying cause for 3.1 million deaths of children younger than 5 years. 18.7 million children under five years of age suffer from severe acute malnutrition (SAM) and an additional 33 million children suffer from moderate acute malnutrition, and are at risk of developing SAM

In Sub-Saharan Africa, there is often poor integration between programs to treat child acute malnutrition and programs that focus on the prevention of acute and chronic undernutrition - resulting in many missed opportunities for using prevention platforms to screen and refer SAM children, or for using screening and referral platforms to provide prevention services.

This project will address two critical gaps related to the integration of preventive and treatment programs: 1) screening and treatment of MAM/SAM have not yet been systematically integrated into routine health-center visits or mainstreamed into community outreach programs; and 2) screening programs often do not offer any preventive services for those children found not to be suffering from MAM/SAM at the time of screening; mothers of children identified as non-MAM/SAM case are usually sent home without receiving any health or nutrition inputs and as a result, may fail to come back for screening because they do not see any tangible benefit associated with their participation in the screening. This project will specifically address these gaps by assessing the effect of an integrated approach consisting of higher screening coverage and preventive Behavior Change Communication (BCC) + Small-Quantity Lipid-based Nutrient supplementation (SQ-LNS) on both prevention and treatment of child undernutrition.

DETAILED DESCRIPTION:
Because of the intended dual role of BCC/SQ-LNS on child undernutrition in this study - e.g. to help prevent child undernutrition and enhance the coverage of screening, referral and treatment of SAM/MAM, it is necessary to combine two study designs to rigorously evaluate the impact of the proposed intervention and to tease out the contribution of prevention and enhanced coverage/treatment to the overall impact on child malnutrition.

The proposed study will therefore use two types of study designs. The first one is a repeated cross-sectional design that will compare select study outcomes between intervention and control groups at endline, after 24 months of program implementation. A repeated cross-sectional study design among children 0-17 months, at baseline and at study endline (on different children) will be used to assess the impact of the intervention on the prevalence of several outcomes, including the prevalence of MAM/SAM and stunting, the coverage of MAM/SAM screening and maternal ENA/IYCF/WASH knowledge and practices. The second proposed study design entails a longitudinal design whereby individual children will be recruited at birth and followed-up monthly until they reach 18 months of age. We anticipate needing approximately 5 months to recruit the required number of children (estimated at 2,040- 1,020 in the control group and 1,020 in the intervention group). This design will allow us to assess the intervention's effects on the incidence, recovery and recurrence rates of MAM/SAM.

ELIGIBILITY:
Cross-sectional study (baseline and endline) (n=2,310)

Inclusion Criteria:

* At least one index child 0-17 months of age in the household
* Mother should be living in the study area since the index child's delivery
* Singleton infants

Exclusion Criteria:

- Index child should not present congenital deformations that hamper anthropometric measurements

Longitudinal study (n=2,180)

Inclusion Criteria:

* child 0-1.4 months of age;
* Mother should be living in the study area since the index child's delivery
* Singleton infants

Exclusion Criteria:

* Congenital malformations that make anthropometric measurements impossible
* Mother planning to leave the study area in the coming year
* Children of 1.5 month of age or older at study inclusion
* WHZ<-2 both at enrollment and at the first follow-up.

Max Age: 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2014-10-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute child malnutrition defined by WHZ<-2 or MUAC <125mm or bilateral pitting edema in children 0-17 months of age | After 24 months of program implementation
  * Cross-sectional study
  * To calculate WHZ scores the 2006 WHO growth reference will be used
  * The MUAC criterion (125mm) is only used for children 6-17months of age
Screening coverage of acute child malnutrition (proportion of children monthly screened / total number of eligible children (aged 0-17 months) | monthly from study inclusion at 0 months to 17 months of age and at study endline
  * Cross-sectional study
  * Longitudinal study
Incidence of child acute malnutrition defined by WHZ<-2 or MUAC<125mm | monthly from study inclusion at 0 months to 17 months of age
  * Longitudinal study
  * To calculate WHZ scores the 2006 WHO growth reference will be used
Compliance to treatment of acute malnutrition (% of cases that complete treatment over total admitted) | monthly from study inclusion at 0 months to 17 months of age and at study endline
  * Cross-sectional study
  * Longitudinal study

SECONDARY OUTCOMES:
Prevalence of child stunting defined by HAZ<-2 in children 0-17 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Mean WHZ-score in children 0 -17 months of age | After 24 months of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Mean HAZ-score in children 0-17 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Mean mid-upper arm circumference in children 0-17 months of age | After 24 months of program implementation
Mean hemoglobin concentration in children 3-17 months of age | After 24 months of program implementation
  Hemocues will be used to measure Hb concentration
Prevalence of child anemia (Hb concentration<10g/dL) in children 3 - 17 months of age | After 24 months of program implementation
Prevalence of severe acute child malnutrition defined by a WHZ<-3 or bilateral pitting edema or a MUAC<115mm in children 0-17 months of age | After 24 months of program implementation
  The MUAC criterion (115mm) is only used for children 6-17months of age
Prevalence of severe stunting defined by a HAZ<-3 in children 0-17 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Caregiver's knowledge and practices related to Infant and Young Child Feeding (IYCF), Essential Nutrition Actions (ENA) and Water, Sanitation and Hygiene (WASH) | After 24 months of program implementation
Incidence of child stunting defined by HAZ<-2 in children from 0 to 17 months | monthly from inclusion at 0 months to 17 months of age
  To calculate HAZ score the 2006 WHO growth reference will be used
Linear growth velocity (HAZ increment/month) | monthly from inclusion at 0 months to 17 months of age
  To calculate HAZ score the 2006 WHO growth reference will be used
Ponderal growth velocity (WHZ increment/month) | monthly from inclusion at 0 months to 17 months of age
  To calculate WHZ score the 2006 WHO growth reference will be used
Weight gain (weight increment/month) | monthly from inclusion at 0 months to 17 months of age
Mid-upper arm circumference gain (MUAC increment/month) | monthly from inclusion at 0 months to 17 moths of age
Infant morbidity (acute respiratory infections, fever, malaria (RDT), vomiting, diarrhea) | monthly from inclusion at 0 months to 17 moths of age
  Malaria will be tested in case of fever (or recalled fever over last 24hrs) use rapid tests
Relapse rate after treatment of MAM/SAM (proportion WHZ<-2 or MUAC<125mm or bilateral pitting edema after discharge from MAM or SAM treatment program over total number of children treated) | monthly from inclusion at 0 months to 17 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ruel, PhD, Principal Investigator — International Food Policy Research Institute; Jean-Celestin Somda, MD, Principal Investigator — Helen Keller International
Locations (1):
- Gourcy Health District, Gourcy, Région Du Nord, Burkina Faso

REFERENCES:
- [Derived] Becquey E, Huybregts L, Zongrone A, Le Port A, Leroy JL, Rawat R, Toure M, Ruel MT. Impact on child acute malnutrition of integrating a preventive nutrition package into facility-based screening for acute malnutrition during well-baby consultation: A cluster-randomized controlled trial in Burkina Faso. PLoS Med. 2019 Aug 27;16(8):e1002877. doi: 10.1371/journal.pmed.1002877. eCollection 2019 Aug. PMID 31454347
- [Derived] Huybregts L, Becquey E, Zongrone A, Le Port A, Khassanova R, Coulibaly L, Leroy JL, Rawat R, Ruel MT. The impact of integrated prevention and treatment on child malnutrition and health: the PROMIS project, a randomized control trial in Burkina Faso and Mali. BMC Public Health. 2017 Mar 9;17(1):237. doi: 10.1186/s12889-017-4146-6. PMID 28274214